CLINICAL TRIAL: NCT04794192
Title: Assessment of the Ankle Systolic Pressure Index in Patients Over 70 Years of Age With Jaundice Ulcer
Acronym: IPScheville
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: IPS cheville
Record Dates: First submitted 2021-03-05; First posted 2021-03-11 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Arteriopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Arteriopathy of the lower limbs (ALL) is defined by a decreased ankle perfusion pressure with a systolic pressure index (SPI) <0.9, and constitutes the most advanced situation in terms of cardiovascular prognosis with in 20 % of cases of lesions associated with the heart and / or coronary heart. The severity of ALL is linked to the risk of a cardiovascular event, hence the need for a hemodynamic evaluation which is mainly based on the measurement of SPI.

DETAILED DESCRIPTION:
However, the presence of mediacalcosis, making the arteries incompressible, limits the interpretation of IPS. However, ALL affects 50% of diabetic patients after 20 years of disease with predominant involvement in the infra-popliteal gland consisting mainly of mediacalcosis, but often respecting the arteries of the foot.

The recommendations of the French-speaking Association for the Study of Diabetes and Metabolic Diseases in 1997 and of the American Diabetes Association in 2001, recommended the SPI and the realization of ultrasound for the diagnosis of ALL. Some authors have shown that SPI can be falsely normal with 4.3 times more false negative ankle SPI in diabetics compared to the general population. This is why this measurement of the SPI is coupled with the measurement of the pressure of the big toe (PGT) or even the transcutaneous measurement of the oxygen pressure (TcPO2) as recommended by the American Heart Association (AHA) and the American College of Cardiology (ACC) in 2005, in case of uninterpretable IPS.

The subjects at risk of mediacalcosis are: diabetics, renal insufficiency and the very elderly.

A recent thesis work confirmed that the SPI alone was not reliable as a screening tool in diabetic patients, with good sensitivity of the measurement of PGT.

What about a population over the age of 70, without diabetes and without kidney failure?

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged> 70 hospitalized in the vascular medicine department of the Paris Saint-Joseph Hospital Group
* French-speaking patient

Exclusion Criteria:

* Patient with treated or untreated diabetes
* Renal failure (GFR CKD-EPI or MDRD <60ml / min)
* ATCD revascularization or amputation
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient objecting to participation in the study
* Patient under legal protection.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged> 70 hospitalized in the vascular medicine department of the Paris Saint-Joseph Hospital Group
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of toe IPSI by laser-doppler, as a screening test for ALL in patients over 70 years of age, non-diabetic and non-renal failure, compared to the data of the considered Doppler ultrasound as the gold standard | Day 1
  Sensitivity and specificity of laser-doppler toe PSI for screening ALL in patients over 70 years of age.

SECONDARY OUTCOMES:
Determination of the age of the population | Day 1
  Age
Determination of the sex of the population | Day 1
  Sex
Number of participants with presence of hypertension | Day 1
  Presence of hypertension
Number of smokers among the participants | Day 1
  Tobacco
Number of participants with cardiovascular history | Day 1
  Cardiovascular history
Number of participants with treatments | Day 1
  Treatments
Relationship between toe SPI and risk factors for arterial disease of the lower limbs | Day 1
  SPI toe values by subgroups of risk factors for arterial disease of the lower limbs
Relationship between ankle SPI and lower limb arterial disease risk factors | Day 1
  SPI ankle values by subgroups of risk factors for arterial disease of the lower limbs
Search for predictive factors associated with toe SPI for the diagnosis of arteriopathy of the lower limbs | Day 1
  Predictors associated with toe PSI for the occurrence of lower limb arterial disease
Search for predictive factors associated with ankle SPI for the diagnosis of arteriopathy of the lower limbs | Day 1
  Predictors associated with ankle PSI for the occurrence of lower limb arterial disease

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël ATTAL, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France